CLINICAL TRIAL: NCT02701764
Title: Can Pregabalin Reduce the Frequency and Severity of Dry Eye Symptoms After Laser-assisted in Situ Keratomileusis?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anat Galor, Associate Professor of Clinical Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20160095
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye
Keywords: laser-assisted in situ keratomileusis; dry eye symptoms; LASIK; prevention
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 150 mg twice a day starting 1 day prior to LASIK and continuing for 14 days total.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo pill twice a day starting 1 day prior to LASIK and continuing for 14 days total.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin
  Arms: Pregabalin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Can Lyrica (Pregabalin) help prevent severe Dry Eye post LASIK surgery?

DETAILED DESCRIPTION:
Dry eye symptoms can occur after LASIK surgery. They generally get better with time but in some patients, they can persist. The investigators believe that in some individuals, dry eye symptoms after LASIK persist because the nerves in the cornea become hypersensitive. The investigators wish to study if a medication, called pregabalin, can protect corneal nerves at the time of LASIK surgery and decrease the frequency and severity of dry eye symptoms 6 months after surgery. This medication has been used in a similar way to reduce the frequency of uncomfortable sensations after other surgeries (knee, abdomen) but has never been studied in LASIK surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years of age
* undergoing LASIK (unilateral or bilateral procedure).
* Females of child-bearing age will need a negative urine or serum pregnancy test at the screening visit.
* ocular and systemic medication regimen has been stable for 3 months

Exclusion Criteria:

* Pregnant or lactating, participating in another study with an investigational drug within one month prior to screening
* Using gabapentin, pregabalin, anti-convulsants, duloxetine, venlafaxine (SNRI), or tri-cyclic antidepressants
* have a history of allergic, anaphylactic reaction, or severe systemic response to pregabalin or gabapentin
* use corticosteroids chronically or during the month prior to surgery, or have a history of corneal disease (HSV or varicella zoster keratitis, prior corneal incisions (cataract surgery, radial keratotomy, LASIK), prior corneal ulcer).
* patients with systemic co-morbidities that may confound DE such as HIV, sarcoidosis, graft-versus host disease or a collagen vascular disease.
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anat Galor, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- Anat Galor, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levitt AE, Galor A, Weiss JS, Felix ER, Martin ER, Patin DJ, Sarantopoulos KD, Levitt RC. Chronic dry eye symptoms after LASIK: parallels and lessons to be learned from other persistent post-operative pain disorders. Mol Pain. 2015 Apr 21;11:21. doi: 10.1186/s12990-015-0020-7. PMID 25896684
- [Derived] Levitt AE, Galor A, Small L, Feuer W, Felix ER. Pain sensitivity and autonomic nervous system parameters as predictors of dry eye symptoms after LASIK. Ocul Surf. 2021 Jan;19:275-281. doi: 10.1016/j.jtos.2020.10.004. Epub 2020 Oct 21. PMID 33096271

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin 150 mg twice a day starting 1 day prior to LASIK and continuing for 14 days total.
  Pregabalin
- Placebo: Placebo pill twice a day starting 1 day prior to LASIK and continuing for 14 days total.
  Placebo
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.8) | 33.0 (0.6) | 35.33 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 7 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Severity of Dry Eye Symptoms as Assessed by the Dry Eye Questionnaire - 5 (DEQ5)
Description: DEQ5 total score ranges from 0-22 with the higher scores indicating increased dry eye. Absolute score will be reported from DEQ5 questionnaire completed at 6 month visit.
Time Frame: 6 months
Population: One participant in the placebo group did not complete 6 month visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 21
score on a scale | 6.6 (5.0) | 4.5 (4.2)

2. Secondary Outcome: Dry Eye Symptoms as Evaluated by the Ocular Surface Disease Index (OSDI)
Description: OSDI total score ranges from 0-100 with a higher score indicating greater disability. Absolute scores will be reported from OSDI questionnaire completed at 3 and 6 month visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  3 months | 11.9 (11.5) | 11.0 (16.6)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 12.6 (15.0) | 12.3 (16.8)

3. Secondary Outcome: Tear Production Measured by Schirmers Score
Description: Tear production will be measured via Schirmers score. Schirmer strips will be placed in the outer 1/3 of the lower conjunctivae. The Schirmer score will be evaluated as the length of wetting in mm in the Schirmer strips after 5 minutes. Absolute scores will be reported for the tear production evaluation at the 3 and 6 months visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit
Measure: Mean (Standard Deviation); unit: mm wetting
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
mm wetting
  3 months | 12.40 (8.71) | 15.90 (9.32)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 15.45 (8.17) | 15.05 (8.64)

4. Secondary Outcome: Tear Evaporation Measured by Tear Break up Time (TBUT)
Description: Participant will have 5 μl of preservative free fluorescein placed on their eye. The participant will then be positioned in the head rest of the slit lamp instrument and will be instructed to blink three times naturally and then not blink. The integrity of the tear film will be measured and, using a stopwatch, the time from the last blink until one or more black (dry) spots appear in the precorneal tear film will be recorded as TBUT. The absolute scores for TBUT completed on the 3 and 6 month visit will be reported.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete 6 month visit
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
Seconds
  3 months | 7.10 (3.87) | 9.54 (5.58)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 8.35 (2.46) | 9.05 (5.93)

5. Secondary Outcome: Eye Pain as Evaluated by the Neuropathic Pain Symptom Inventory - Eye (NPSI-E)
Description: NPSI-E total score ranges from 0-100 with a higher score indicating increased eye pain. Absolute scores will be reported from NPSI-Eye questionnaire completed at 3 and 6 month visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  3 months | 2.70 (4.55) | 1.86 (4.07)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 2.81 (4.07) | 3.14 (5.85)

6. Secondary Outcome: Eye Pain as Assessed by the Short Form - McGill Pain Questionnaire (Sf-MPQ) Sensory
Description: sf-MPQ Sensory has a total score ranging from 0-33 with a higher score indicating increased pain. Absolute scores will be reported from sf-MPQ Sensory questionnaire completed at 3 and 6 month visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  3 months | 0.65 (1.23) | 0.36 (0.66)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 0.48 (1.03) | 0.81 (2.42)

7. Secondary Outcome: Eye Pain as Assessed by the Short Form - McGill Pain Questionnaire (Sf-MPQ) Affective
Description: sf-MPQ Affective has a total score ranging from 0-12 with a higher score indicating increased pain. Absolute scores will be reported from sf-MPQ Affective questionnaire completed at 3 and 6 month visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  3 months | 0.30 (0.66) | 0.18 (0.39)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 0.29 (0.46) | 0.43 (0.98)

8. Secondary Outcome: Eye Pain as Assessed by the Numeric Rating Scale (NRS)
Description: NRS total score ranges from 0-10 over a one week recall period with the higher score indicating increased pain. Absolute scores will be reported from NRS questionnaire completed at 3 and 6 month visit.
Time Frame: 3 months, 6 months
Population: One participant in the placebo group did not complete the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  3 months | 0.85 (0.27) | 0.27 (0.55)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 1.10 (1.48) | 0.38 (0.97)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pregabalin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 13/21 | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=21) | Placebo (N=22)
Tiredness (General disorders) | 8 | 2
Dizziness (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Bloating (Gastrointestinal disorders) | 3 | 4
High or elevated mood (Psychiatric disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT02701764/Prot_SAP_000.pdf